CLINICAL TRIAL: NCT03114774
Title: Evaluation of Effectivity of Bispectral Index Monitoring in Cases of Endoscopic Retrograde Cholangiopancreatography Received Sedoanalgesia
Brief Title: Effectivity of Bispectral Index Monitoring in Cases of Endoscopic Retrograde Cholangiopancreatography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ferda Yilmaz Inal, Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 71306642-050.01.04-21/29
Record Dates: First submitted 2017-03-20; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Sedoanalgesia
MeSH Terms: interventions — GRB10 Adaptor Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grup 1: Ramsay Sedation Scale (RSS) Score monitoring
  Interventions: Behavioral: Ramsay Sedation Scale (RSS) Score monitoring
- Grup 2: The bispectral index (BIS) monitoring
  Interventions: Device: The bispectral index (BIS) monitoring

INTERVENTIONS:
Device: The bispectral index (BIS) monitoring
  Groups: Grup 2
Behavioral: Ramsay Sedation Scale (RSS) Score monitoring
  Groups: grup 1

SUMMARY:
The bispectral index (BIS) monitoring is an EEG-based method that uses electroencephalogram analysis and a complex algorithm to generate a numerical scoring 0-100 (0 flat line EEG, 100, wide awake) BIS monitoring allows noninvasive, objective measurement of level of consciousness of a sedated patient. A limited number of studies have used measurements of BIS monitoring to assist endoscopic sedation.There are studies using BIS monitoring to make sedation easy for ERCP procedures. However, the studies evaluating use of BIS for gastrointestinal endoscopy show inconsistent results.

The objective of this study is to evaluate effects of sedation on the dosage of propofol by monitoring with BIS values, hemodynamics, recovery parameters, respiratory functions and endoscopist satisfaction based on the hypothesis that the investigators would reduce the risk for respiratory depression using minimal doses of propofol in order to achieve the desired level of sedation with BIS monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75 years old
2. ASA 1-2

Exclusion Criteria:

1. Emergency Operation
2. Those who had symptoms of neurological disease (TİA, syncope, dementia, etc.)
3. Patients that are allergic to drugs considered to use

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients in ASA 1-2 category scheduled for sedation and ERCP
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-06-01 (Estimated)

PRIMARY OUTCOMES:
Total dosage of propofol | 1-3 hours
  initial dose 1 mg.kg-1 of propofol, maintenance dose: infusion of 4 mg/kg/h . In case of insufficient sedation, additional dose of 0.1 mg/kg propofol (IV) by monitoring with BIS values 65-75 during procedure
The heart rate (HR)(n/dk) | 1-3 hours
  During procedure
mean systolic-diastolic blood pressure(mmHg) | 1-3 hours
  during procedure
peripheral oxygen saturation (%) | 1-3 hours
  During procedure